CLINICAL TRIAL: NCT01135641
Title: Phase II Study of First Line Treatment of Chronic Graft Versus Host Disease With the Association of Ciclosporine, Corticosteroids and Rituximab
Brief Title: Study of First Line Treatment of Chronic Graft Versus Host Disease With the Association of Ciclosporine, Corticosteroids and Rituximab (Protocol R-GVHD)
Acronym: R-GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/6-B; 2009-016898-14 (EudraCT Number)
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Graft Versus Host Disease
Keywords: Adult patients (≥18 years); first allogeneic stem cell transplantation; first episode of chronic GVHD requiring systemic immunosuppressive therapy
MeSH Terms: conditions — Graft vs Host Disease | interventions — Rituximab; Cyclosporins; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab, ciclosporine and corticosteroids (Experimental): As soon as the diagnosis of chronic GVHD requiring systemic immunosuppressive therapy is confirmed, patients will receive in addition to ciclosporine A and corticosteroids (prednisone) 1 mg/kg/day, Rituximab at 375 mg/m²/infusion once a week for 4 consecutive weeks.Rituximab should be administered within 14 days of starting prednisone. Follow-up dates for response assessment and laboratory tests relate to the date of Rituximab infusion.Patients having a partial response after the 1st cycle of Rituximab will be eligible to receive a second cycle of 4 infusions during 4 weeks. A delay of 8 weeks (from the first infusion of Rituximab) will be observed between the two cycles of Rituximab therapy.Patients who relapse after an initial treatment with one cycle of 4 infusions of Rituximab will be eligible to receive a second cycle of Rituximab therapy.
  Interventions: Drug: Rituximab; Drug: Ciclosporine; Drug: Corticosteroids

INTERVENTIONS:
Drug: Rituximab — Patients will receive in addition to ciclosporine A and corticosteroids (prednisone) 1 mg/kg/day, Rituximab at 375 mg/m²/infusion once a week for 4 consecutive weeks.
Drug: Ciclosporine
Drug: Corticosteroids

SUMMARY:
The main objective of the study is to improve the response rate (complete and partial remission) at 12 months after diagnosis of chronic Chronic Graft Versus Host Disease (GVHD) and treatment with the combination of ciclosporine, prednisone and Rituximab as first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who have received a first allogeneic stem cell transplantation for a hematological disease
* Confirmed diagnosis of first episode of chronic GVHD requiring systemic immunosuppressive therapy. Chronic GVHD diagnosis is defined according to the NIH Working Group Consensus. Chronic GVHD diagnosis will be based on the evaluation of the severity of the different clinical manifestations including :

  1. Ocular, oral and mucosal symptoms,
  2. Performance status evaluation,
  3. Pulmonary function evaluation,
  4. Cutaneous evaluation measured by the percentage of extension of manifestations of liche-noid or sclerodermatous aspects, eventually confirmed with a biopsy whenever possible,
  5. Evaluation of the musculoskeletal manifestations, especially the amplitude of the rele-vant articulations,
  6. Evaluation of liver involvement (Total bilirubin, Transaminases, Phosphatase alcalines and Gamma GT).
* Any source of hematopoietic stem cells is authorized.
* Any category of conditioning regimen prior to allo-SCT is authorized.
* Any type of stem cell donors is authorized.
* Signed informed consent.
* Any prior GVHD prophylaxis previously used is accepted.
* Absence of contra-indications to the use of Rituximab.
* Subjects affiliated with an appropriate social security system.
* Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception throughout the study and for 3 months following the end of the study.

Exclusion Criteria:

* Patient developing acute GVHD (whether early or "late onset" form)
* A "limited" form of chronic GVHD not requiring systemic immunosuppressive therapy
* Treatment with prednisone (or equivalent) at doses higher than 1 mg/kg/day at the time of enrollment.
* GVHD occurring following donor lymphocytes infusion (DLI)
* Not the first episode of chronic GVHD needing systemic immunosuppressive therapy
* Neutropenia <500/µL
* Second allogeneic stem cell transplant
* Uncontrolled systemic infection which in the opinion of the investigator is associated with an increased risk of the patient's death within 1 month after the start of therapy
* Severe neurological or psychiatric disorders
* Denied informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response rate at 12 months
  Response rate (complete and partial remission) at 12 months after diagnosis of chronic GVHD and treatment with the combination of ciclosporine, prednisone and Rituximab as first line treatment.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability
  To spare patients from long-term use of corticosteroids (and of their long-term side effects)
Treatment failure
  To document treatment failure-defined as initiation of another immunosuppressive agent
Transplant-related mortality
  To decrease transplant-related mortality (TRM) of infectious and non-infectious origin
Quality of life
  To improve quality of life parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, Profesor, Principal Investigator — Hôpital Saint-Antoine (Paris); Noël MILPIED, Profesor, Study Chair — University Hospital, Bordeaux; Mauricette MICHALLET, Profesor, Study Chair — Hospices Civils de Lyon; Karin BILGER, Doctor, Study Chair — CHRU de Strasbourg; Oumédaly REMAN, Doctor, Study Chair — CHRU de Caen; Ibrahim YAKOUB-AGHA, Profesor, Study Chair — CHRU de Lille; Didier BLAISE, Profesor, Study Chair — Institut Paoli-Calmettes; Patrice CEBALLOS, Doctor, Study Chair — CHU de Montpellier; Patrice CHEVALLIER, Doctor, Study Chair — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Malard F, Labopin M, Yakoub-Agha I, Chantepie S, Guillaume T, Blaise D, Tabrizi R, Magro L, Vanhove B, Blancho G, Moreau P, Gaugler B, Chevallier P, Mohty M. Rituximab-based first-line treatment of cGVHD after allogeneic SCT: results of a phase 2 study. Blood. 2017 Nov 16;130(20):2186-2195. doi: 10.1182/blood-2017-05-786137. Epub 2017 Sep 1. PMID 28864814